CLINICAL TRIAL: NCT00975442
Title: Effects of Eccentric Training for Patients With Lateral Epicondylalgia - a Randomized Controlled Trial
Brief Title: Effects of Eccentric Training for Patients With Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Rehband Sweden (Unknown)
Responsible Party: Johan Söderberg P.T., Department of Neurobiology, Care Sciences and Society, Division of Physiotherapy, Karolinska Institutet, Huddinge, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 221/00
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Tennis Elbow; Epicondylitis, Lateral Humeral
Keywords: Elbow; Tendinitis; Sports Medicine; Athletic injuries
MeSH Terms: conditions — Tennis Elbow; Tendinopathy; Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric training (Experimental)
  Interventions: Other: Eccentric training; Device: Forearm band
- Forearm band (Placebo Comparator)
  Interventions: Device: Forearm band

INTERVENTIONS:
Other: Eccentric training — A home training program of eccentric training of the wrist extensors to be carried out daily with 3 sets of 15 repetitions. All subjects were instructed to use the forearm band (Epi Forsa 4061, Rehband, Sweden)
  Arms: Eccentric training
Device: Forearm band — All subjects were instructed to use the forearm band during all daily activities.
  Other Names: Epi Forsa 4061, Rehband, Sweden
  Arms: Forearm band
Device: Forearm band — All patients were instructed to use a forearm band during all daily activities.
  Other Names: Epi Forsa 4061, Rehband, Sweden
  Arms: Eccentric training

SUMMARY:
The purpose of this study is to evaluate eccentric training as an intervention for lateral epicondylalgia (tennis elbow) in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic criteria according to Haker (1991): A history of pain around the lateral epicondyle for at least one month.
* Pain at palpation of the lateral epicondyle of humerus and positive results in two of the following three pain provocation tests: Middle finger test, resisted extension of the wrist, and Vigorimeter test. Each of these tests is described in detail by Haker (1991)

Exclusion Criteria:

* Subjects with rheumatoid arthritis
* Fibromyalgia
* Previous surgery in the elbow region
* Neck dysfunction suggesting possible cervical rhizopathy
* Entrapment of n.radialis
* Patients with ongoing treatment, or previous treatment less than three months before enrolled to the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic criteria, whether or not the patient had recovered according to the diagnostic criteria for LE, Haker (1991) at follow up examinations | 3 wk and 6 wk follow up

SECONDARY OUTCOMES:
Measurements of pain free functional grip strength using the Martin Vigorimeter test, and maximum pain free isometric extensor strength by using Nicholas Myometer | 3 wk and 6 wk follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Johan Söderberg, P.T., Principal Investigator — Department of Neurobiology, Care Sciences and Society, Division of Physiotherapy, Karolinska Institutet, Huddinge, Sweden
Locations (1):
- Karolinska Institutet, Stockholm, Sweden